CLINICAL TRIAL: NCT02242500
Title: Phase IV Study of Coronally Advanced Flap With or Without Porcine Collagen Matrix for Treatment of Gingival Recession: a Randomized Controlled Clinical Trial
Brief Title: Coronally Advanced Flap With or Without Porcine Collagen Matrix for Root Coverage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Enilson Antonio Sallum (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor-Investigator, Enilson Antonio Sallum, Chair of the Department of Prosthodontics and Periodontics, Division of Periodontics, Piracicaba Dental School, University of Campinas, Brazil
Organization: University of Campinas, Brazil (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 130/2010
Record Dates: First submitted 2014-09-13; First posted 2014-09-17 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Gingival Recession
Keywords: Gingival recession/surgery; Collagen/therapeutic use; Root coverage; Treatment outcome
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coronally advanced flap + Mucograft (Experimental): coronally advanced flap associated with a porcine collagen matrix graft as a subepithelial graft
  Interventions: Procedure: Coronally Advanced Flap; Device: Mucograft
- Coronally advanced flap (Other): Coronally advanced flap procedure alone
  Interventions: Procedure: Coronally Advanced Flap

INTERVENTIONS:
Procedure: Coronally Advanced Flap
Device: Mucograft
  Other Names: Porcine collagen matrix for soft tissue regeneration
  Arms: Coronally advanced flap + Mucograft

SUMMARY:
The purpose of this study is to compare the clinical outcomes after coronally advanced flap technique (CAF) associated or not to a porcine collagen matrix graft (CM) in the treatment of single gingival recessions. For this blinded randomized controlled clinical trial, 40 patients with Miller Class I or II gingival recession ≥ 2 mm in canines or premolars will selected and randomly assigned to receive either CAF or CAF+CM. The clinical parameters evaluated will be probing depth, clinical attachment level, gingival recession height, height and thickness of keratinized tissue. Clinical measurements will be taken at baseline and 45 days, 2, 3 and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Presence of at least one Class I or II Miller gingival recession ≥ 2 mm in maxillary canines or premolars with identifiable cementum-enamel junction (CEJ) and without deep non-carious cervical lesions (< 0.5 mm): A + (Pini-Prato et al. 2010).
* Aesthetic complaint and/or presence of dentin hypersensitivity to air stimulus.
* Full-mouth visible plaque index ≤ 20% (Ainamo & Bay 1975).
* Full-mouth sulcus bleeding index ≤ 20% (Mühlemann & Son 1971).

Exclusion Criteria:

* Smoking.
* Pregnancy.
* Presence of systemic disorders (diabetes, hypertension, heart disease or any other condition that could contraindicate periodontal surgery).
* Use of medications (immunosuppressants, phenytoin or anything else that might affect mucosal healing and repair).
* Previous periodontal surgery in the area.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Recession Reduction | 6 months
  Measured as a difference between gingival margin between gingival recession depth at baseline and gingival recession at 6 months follow-up.

SECONDARY OUTCOMES:
Complete root coverage | 6 months
  Assessed as percentage of sites with complete root coverage

OTHER OUTCOMES:
Keratinized tissue thickness | 6 months
  Measured at a midpoint between gingival margin and mucogingival junction using a endodontic spreader pierced perpendicular and through the soft tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Piracicaba Dental School, State University of Campinas, Piracicaba, São Paulo, Brazil